CLINICAL TRIAL: NCT06658041
Title: Effectiveness of a Collaborative Stepped-care Intervention for Adults Aged 45 and Above With Subthreshold Depressive Symptoms in the Primary Care Setting in Hong Kong
Brief Title: Collaborative Stepped-care Intervention for Adults With Subthreshold Depressive Symptoms in the Primary Care Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Baptist Oi Kwan Social Service (Other); Caritas Medical Centre, Hong Kong (Other); Christian Family Service Centre (Other); Fu Hong Society (Unknown); Haven of Hope Hospital (Other); Hong Kong Christian Service (Other); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Young Women's Christian Association (Other); The Mental Health Association of Hong Kong (Other); Neighbourhood Advice-Action Council (Other); New Life Psychiatric Rehabilitation Association (Other); Richmond Fellowship of Hong Kong (Unknown); Hong Kong Sheng Kung Hui Lady MacLehose Centre (Unknown); SideBySide (Unknown); St. James' Settlement (Other); The Hong Kong Society for the Aged (Unknown); The Salvation Army, Hong Kong and Macau Command (Other); Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-246
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Depressive symptoms; Mental health; Primary care; Stepped-care intervention
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Cognitive Behavioral Therapy; Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: A quasi-experimental randomised controlled trial with propensity score-matching of an (i) intervention arm and (ii) active control arm.
Masking Description: Masking was not possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JoyAge stepped-care intervention (Experimental): Participants are provided with specified interventions (cognitive behavioural therapy-based) according to their depressive symptom severity at the primary care setting provided by trained clinical social workers, and may be stepped-up or stepped-down according to their response.
  Interventions: Behavioral: Cognitive behavioural therapy (CBT)-based intervention with stepped-care
- Care-as-usual (Active Comparator): Participants will continue with any services they are receiving (non-JoyAge intervention), which may entail services such as stress management or health-related programmes but without symptom-specific psychological interventions or stepped-care.
  Interventions: Other: Care-as-usual

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy (CBT)-based intervention with stepped-care — After initial clinical assessment, participants will be offered interventions based on their depressive symptom severity (Patient Health Questionnaire-9-item [PHQ-9]).
  Mild symptoms (PHQ-9=5-9) without major risks (*see above): 4 weekly CBT-informed intervention sessions led by trained Emotional Support Assistants (Peer Supporters with 80hrs mental health training + 15hrs intensive clinical training).
  Mild symptoms (PHQ-9=5-9) with major risk factors or moderate-to-moderately severe symptoms (PHQ-9=10-19): 6 weekly CBT-based intervention sessions led by trained clinical social workers, with 2 booster sessions as necessary. Individual CBT-based intervention will be provided to those unsuitable for group interventions.
  In cases of non-remission (PHQ-9≥5): a second intervention trial will be provided. Those needing additional support will be referred to a partnered General Practitioner (if PHQ-9=10-19) or referred to more intensive psychological or psychiatric services as needed.
  Other Names: Psychological intervention; Stepped-care intervention
  Arms: JoyAge stepped-care intervention
Other: Care-as-usual — Following an initial interview session with research assessments, participants continue with their usual care at their primary care setting.
  Other Names: CAU
  Arms: Care-as-usual

SUMMARY:
To ensure accessibility and availability of mental health services in the community and to reduce the burden associated with depression and related conditions, the study aim to evaluate the effectiveness of a collaborative stepped-care intervention (cognitive behavioural therapy-based) for adults with subthreshold depressive symptoms at the district-based primary healthcare setting.

DETAILED DESCRIPTION:
Depression is among the most prevalent mental health conditions globally and contributes substantially to the global burden of disease. In adults, depression is highly comorbid not only with other mental health conditions (e.g., anxiety) but also physical diseases.

Since 2016, the research team has developed a collaborative stepped-care model for older people at-risk of or with depression in Hong Kong through the Jockey Club Holistic Support Project for Elderly Mental Wellness (JC JoyAge) (Clinical Trials Identifier: NCT03593889); the effectiveness and cost-effectiveness of which has been demonstrated, thereby leading to its implementation in social care settings across all 18 districts of Hong Kong.

To further improve the accessibility and availability of mental health services in the community and to reduce the burden associated with depression and related conditions, the JoyAge collaborative stepped-care intervention (cognitive behavioural therapy-based) will be expanded to target adults aged 45 years and above at the district-based primary care setting. This study thus sought to evaluate the effectiveness of this expanded intervention model.

Objective: To examine the effectiveness of the collaborative stepped-care intervention for adults with subthreshold depressive symptoms, as compared with propensity score-matched controls, in reducing depressive symptoms (primary outcome) both post-intervention (T1) and for up to 3 months of follow-up (T2). Secondary outcomes of the study include reduced anxiety symptoms, reduced loneliness, reduced rumination, improved social support, improved health-related quality of life, as well as improved quality-adjusted life years, and reduced healthcare service utilisation.

Design: While a randomised controlled trial would be ideal, such a study design was not possible in our current study context given pragmatic reasons. A quasi-experimental randomised controlled trial involving an (i) intervention arm and (ii) control arm will therefore be adopted. A targeted sample of 352 participants will be recruited (n = 176 per arm). To more rigorously account for potential differences in the sample characteristics of the two arms, propensity-score matching will be applied. After the pre-intervention or baseline (T0), assessments will be conducted at two follow-up time points: post-intervention (9-month post-baseline in the active control group, which is aligned with the median service duration in the intervention arm; T1), and 3-month post-intervention (12-month post-baseline in the active control group; T2).

Study setting

In Hong Kong, there is now at least one core district-based primary care centre at each of the 18 districts locally. Aside from the regular JoyAge intervention offered in the social care setting, the present study will focus on the effectiveness of the JoyAge intervention carried out at three main primary care centre sites in Hong Kong. Participants of the control group will be recruited from the community, comprising individuals who may be receiving services from non-JoyAge-partnered district-based primary care centres (that are not actively offering psychological interventions) or other services.

Power calculation for sample size

Taking a more conservative effect size reported in a meta-analysis examining the effects of psychotherapy for subclinical depression (using the lower confidence interval [CI] of CBT, yielding f = 0.14) (Cuijpers et al., 2014), a minimum sample size of 270 is required to achieve a power of 80% at the 0.05 alpha level. Further accounting for a potential 30% attrition given the setting in which this study is conducted, a total sample of 352 is targeted (n = 176 per arm).

Procedures and intervention: Experimental group

For those in the JoyAge partnered district-based primary care centres, participants identified to be showing some symptoms of depression (Patient Health Questionnaire-2-item ≥ 3) will be directed to the JoyAge team for a more in-depth assessment, involving the completion of a full Patient Health Questionnaire-9-item (PHQ-9). Those meeting the study inclusion criteria (see below) and have provided informed consent will be provided with interventions according to initial symptom severity, which are predominantly based on cognitive behavioural therapy (CBT) with a stepped-care element. Details are as follows:

* For those with mild symptoms (PHQ-9 = 5-9) without major risks: 4 weekly CBT-informed intervention sessions led by trained Emotional Support Assistants (ESA) (Peer Supporters with 80hrs mental health training + 15hrs intensive clinical training).
* For those with mild symptoms (PHQ-9 = 5-9) with major risk factors or moderate-to-moderately severe symptoms (PHQ-9 = 10-19): 6 weekly CBT-based intervention sessions led by trained clinical social workers, with 2 booster sessions as necessary. Individual CBT-based intervention will be provided to those unsuitable for group interventions.

Based on the initial trial of intervention, participants may be either "stepped-up" or "stepped-down" (or exit from service). Specifically:

- For all participants who were unable to achieve clinical remission following the first trial of intervention (PHQ-9 ≥ 5): a second trial of intervention will be provided with greater intensity (e.g., those receiving ESA-led interventions may be stepped up to worker-led interventions). Those needing additional support will be referred to a partnered General Practitioner (if PHQ-9=10-19) or referred to more intensive psychological or psychiatric services as needed.

*Definition of major risk factors: PHQ-9 item 9 (suicidal ideation) ≥ 2; moderate symptoms of generalised anxiety disorder (GAD-7 ≥ 10); high loneliness (UCLA 3-item ≥ 7); recent highly stressful or traumatic event (e.g., bereavement, domestic violence); complex high-risk condition (e.g., major family issues).

The recommended service period will be 6-9 months. All assessments will be conducted pre-intervention/baseline (T0), post-intervention (i.e., exit from service; T1), and 3-month post-intervention (T2).

Procedures and intervention: Active control group

Participants will be from community members who are not receiving services from the JoyAge-partnered district-based primary care centres. Upon identification of potential presentation of depressive symptoms, a trained research assistant will further verify their eligibility. Upon confirmation of their eligibility and informed consent provision, assessments will be conducted by a trained research assistant at baseline (T0), at 9-month follow-up (T1) [*aligned with the median service duration in the experimental group], and 12-month follow-up (T2). To ensure the baseline characteristics of the two groups are similar, propensity score matching will be applied, accounting for core demographics (e.g., sex, age) and initial symptom severity (e.g., mild / moderate / moderately severe).

Statistical methods

Sample characteristics will be examined and reported for both experimental arms at all time points. The primary analysis will follow an intention-to-treat (ITT) principle (i.e., all participants will be included as long as they were randomised, and based on their randomised allocation, regardless of the intervention they received or rate of completion).

To test the effects of the intervention on the primary and secondary outcomes of the present study, two approaches will be adopted:

1. Between-group differences will first be analysed using the generalised linear models. Core sociodemographics would be adjusted in these models. Unstandardised coefficients and effect sizes (Cohen's d) with 95% confidence intervals will be reported.
2. Linear mixed models will be applied to further confirm the results, which would account for the random effects at individual participant level.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Hong Kong;
* Presenting mild to moderately severe depressive symptoms (PHQ-9 = 5-19);
* Able to give informed consent to participate.

Exclusion Criteria:

* A known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia;
* Imminent suicidal risk;
* Difficulty in communication that would limit meaningful participation in psychological intervention.

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  The Patient Health Questionnaire-9-item (PHQ-9) is a well-validated measure of depressive symptoms, with items corresponding to the DSM-IV criteria for major depression and which also map onto those of the DSM-V. Items are rated on a 4-point Likert scale and are summed to generate a total score that ranges from 0 to 27. A higher score reflects more severe symptoms.

SECONDARY OUTCOMES:
Changes in anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  The Generalized Anxiety Disorder-7-item (GAD-7) is a well-validated measure of anxiety symptoms, with items also corresponding to symptoms of the DSM. Items are rated on a 4-point Likert scale and are summed to generate a total score that ranges from 0 to 21. A higher score reflects more severe symptoms.
Changes in loneliness symptoms (UCLA Loneliness 3-item [UCLA-3]) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  The UCLA Loneliness 3-item scale (UCLA-3) is a 3-item self-report scale capturing core loneliness experiences, including feeling of a lack of companionship, left out, and isolated. Each item is rated on a 4-point Likert scale, with items summed to generate a total score that ranges from 0 to 9. A higher score reflects higher levels of loneliness.
Changes in depressive rumination (RRS-Brooding) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  The Ruminative Response Scale (RRS) is a commonly used measure for depressive rumination. The brooding subscale is used in particular (RRS-Brooding), which has been shown to be more predictive of poorer outcomes. The RRS-Brooding subscale comprises 5 items assessed on a 4-point Likert scale and are summed to generate a total score that ranges from 5 to 20. A higher score reflects more depressive rumination.
Changes in social network (LSNS-6) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  The 6-item Lubben Social Network Scale (LSNS-6) will be used to assess the self-reported social engagements with family and friends. In this measure, three items are used to examine the social engagements with family and friends, respectively. Each item is rated on a 5-point scale (from "none" to "nine or more" for number of relatives/friends available for each specified social interaction) and are summed to generate a total score that ranges from 0 to 30. A higher score reflects more social engagements.
Changes in health-related quality of life (EQ-5D) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  Health-related quality of life (HR-QoL) will be assessed using the EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L). The EQ-5D-5L is a generic preference-based measure of five core dimensions of health (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels (5L) of problems ranging from 1 to 5, respectively. Results will be presented in the form of EQ-5D-5L index value. The EQ-5D-5L will also be used to calculate quality-adjusted life years.
Changes in service utilisation (CSRI) | T0 (before intervention/baseline); T1 (Intervention group: immediately after intervention; Active control group: 9 months after T0); T2 (3 months after T1)
  Service utilisation will be assessed using the Client Service Receipt Inventory (CSRI) with some adaptations to capture the frequency of service use across different local social and primary care settings.

CONTACTS AND LOCATIONS:
Overall Officials: Terry YS Lum, Ph.D., Principal Investigator — The University of Hong Kong; Gloria HY Wong, Ph.D., Principal Investigator — University of Reading; The University of Hong Kong; Wai Chi Chan, MBChB, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, HONG KONG, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to participant confidentiality reasons.